CLINICAL TRIAL: NCT05582577
Title: Additional Effect of Sub-threshold Micro-pulse Laser to Intra-vitreous Injection of Bevacizumab on Diabetic Macular Edema: A Randomized Double-blinded Clinical Trial
Brief Title: Additional Effect of Subthreshold Micropulse Laser to Intravitreous Injection of Bevacizumab on Diabetic Macular Edema
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of Ophthalmic Research Center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14016
Record Dates: First submitted 2022-09-10; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simultaneous intravitreal bevacizumab injection with subthreshold micropulse laser (Experimental): After the eye examination, the eyes will be randomly divided into 2 groups {group A: intravitreal interjection of Bevacizumab and subthreshold micropulse laser, and group B: intravitreal injection of Bevacizumab alone}. For both groups, 3 intravitreal injections of bevacizumab with a dose of 1.25 mg will be performed, in sterile conditions at 1-month intervals as a loading dose.
  A subthreshold micropulse laser will be performed after the third injection in group A. Then, the intravitreal injection of Bevacizumab will be continued if the central thickness of the macula is equal to or greater than 300 microns.
  The follow-up will be performed 2, 3, 4, 6, 8, 10, and 12 months after the first injection. In each follow-up (except for the first month), ophthalmological examinations and Optical Coherence Tomography will be performed.
  Interventions: Combination Product: Intravitreal bevacizumab injection with subthreshold micropulse laser
- Intravitreal bevacizumab injection alone (Active Comparator): After the eye examination, the eyes will be randomly divided into 2 groups {group A: intravitreal interjection of Bevacizumab and subthreshold micropulse laser, and group B: intravitreal injection of Bevacizumab alone}. For both groups, 3 intravitreal injections of bevacizumab with a dose of 1.25 mg will be performed, in sterile conditions at 1-month intervals as a loading dose.
  A sham laser will be performed after the third injection in group B. Then, the intravitreal injection of Bevacizumab will be continued if the central thickness of the macula is equal to or greater than 300 microns.
  The follow-up will be performed 2, 3, 4, 6, 8, 10, and 12 months after the first injection. In each follow-up (except for the first month), ophthalmological examinations and Optical Coherence Tomography will be performed.
  Interventions: Drug: Intravitreal bevacizumab injection alone

INTERVENTIONS:
Combination Product: Intravitreal bevacizumab injection with subthreshold micropulse laser — Group A: intravitreal interjection of Bevacizumab and subthreshold micropulse laser
  Arms: Simultaneous intravitreal bevacizumab injection with subthreshold micropulse laser
Drug: Intravitreal bevacizumab injection alone — Group B: Intravitreal injection of Bevacizumab alone
  Arms: Intravitreal bevacizumab injection alone

SUMMARY:
In this study, all eyes with diabetic macular edema who meet the inclusion criteria and do not meet the exclusion criteria will be included. After the eye examination, the eyes will be randomly divided into 2 groups {group A: intravitreal interjection of Bevacizumab and subthreshold micropulse laser, and group B: intravitreal injection of Bevacizumab alone}. For both groups, 3 intravitreal injections of bevacizumab with a dose of 1.25 mg will be performed, in sterile conditions at 1-month intervals as a loading dose.

A subthreshold micropulse laser will be performed after the third injection in group A and a sham laser will be performed after the third injection in group B. Then, the intravitreal injection of Bevacizumab will be continued if the central thickness of the macula is equal to or greater than 300 microns.

The follow-up will be performed 2, 3, 4, 6, 8, 10, and 12 months after the first injection. In each follow-up (except for the first month), ophthalmological examinations and Optical Coherence Tomography will be performed.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years diabetic patients
* Center-involved diabetic macular edema
* Mean central subfield thickness >300 micrometers
* Best-corrected visual acuity between 20/40 and 20/400

Exclusion Criteria:

* hemoglobin A1c > 8
* High-risk proliferative diabetic retinopathy
* Prior treatment with intravitreal or peribulbar injections within the preceding 3 months
* History of panretinal photocoagulation within the former 4 months
* History of macular photocoagulation
* Hx of Intraocular surgery (except cataract extraction)
* cataract extraction less than 6 months ago
* Macular edema due to a cause other than diabetic retinopathy
* Any other ocular condition that visual acuity would not improve from the resolution of the edema (eg, foveal atrophy)
* Substantial cataract estimated to have reduced visual acuity by >3 lines
* uveitis, neovascular glaucoma, exudative age-related macular degeneration, high risk proliferative diabetic retinopathy
* vitreomacular traction or epiretinal membrane
* uncontrolled glaucoma ( > 30 millimeters of mercury with anti-glaucoma medications)
* Not having: Media clarity, pupillary dilation, and subject cooperation sufficient for adequate fundus photographs

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline central macular thickness at 2 months | Change from baseline to 2 months
  Change from baseline central macular thickness at 2 months using Optical Coherence Tomography
Change from 2 months central macular thickness at 3 months | Change from 2 months to 3 months
  Change from 2 months central macular thickness at 3 months using Optical Coherence Tomography
Change from 3 months central macular thickness at 4 months | Change from 3 months to 4 months
  Change from 3 months central macular thickness at 4 months using Optical Coherence Tomography
Change from 4 months central macular thickness at 6 months | Change from 4 months to 6 months
  Change from 4 months central macular thickness at 6 months using Optical Coherence Tomography
Change from 6 months central macular thickness at 8 months | Change from 6 months to 8 months
  Change from 6 months central macular thickness at 8 months using Optical Coherence Tomography
Change from 8 months central macular thickness at 10 months | Change from 8 months to 10 months
  Change from 8 months central macular thickness at 10 months using Optical Coherence Tomography
Change from 10 months central macular thickness at 12 months | Change from 10 months to 12 months
  Change from 10 months central macular thickness at 12 months using Optical Coherence Tomography

SECONDARY OUTCOMES:
Change from baseline visual acuity at 2 months | Change from baseline to 2 months
  Change from baseline best-corrected visual acuity at 2 months
Change from 2 months visual acuity at 3 months | Change from 2 months to 3 months
  Change from 2 months best-corrected visual acuity at 3 months
Change from 3 months visual acuity at 4 months | Change from 3 months to 4 months
  Change from 3 months best-corrected visual acuity at 4 months
Change from 4 months visual acuity at 6 months | Change from 4 months to 6 months
  Change from 4 months best-corrected visual acuity at 6 months
Change from 6 months visual acuity at 8 months | Change from 6 months to 8 months
  Change from 6 months best-corrected visual acuity at 8 month
Change from 8 months visual acuity at 10 months | Change from 8 months to 10 months
  Change from 8 months best-corrected visual acuity at 10 months
Change from 10 months visual acuity at 12 months | Change from 10 months to 12 months
  Change from 10 months best-corrected visual acuity at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Ramezani, Principal Investigator — Ophthalmic Research Center, Shahid Beheshti University of Medical Sciences
Locations (1):
- Ophthalmic Research Center, Tehran, Iran